CLINICAL TRIAL: NCT02942511
Title: Predictors Favoring the Role of Exclusive Enteral Nutrition in Active Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, chenyan, Yan Chen, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: SAHZU-GI1
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Crohn's Disease; Enteral Nutrition
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To idetify the factors favoring the use of enteral nutrition would be helpful to select preferred patients suitable for enteral nutrition.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic, transmural inflammatory disorder affecting the whole alimentary tract from mouth to anus. Over the past decades, the incidence of CD is either high and stable or low but rising in the worldwide. Although the precise etiopathogenesis of CD remains unknown, a number of lines of evidence showed that inappropriate diet was one of the reasons responsible for the onset of CD, and diet therapy has been gaining increasing attention in the therapeutic work-up of CD.

Due to reduced intake and high intestinal losses, over three quarters of CD patients would suffer weight loss. Involvement of small bowel in CD patients made their nutrition status much poorer than ulcerative colitis (UC) patients. Therefore, nutrition support is of great value in the management of CD. It is widely accepted that enteral nutrition could help pediatric CD patients to reach clinical and endoscopic remission, with similar efficacy but less side effects than corticosteroids. However, the value of enteral nutrition in adult active CD is still controversial, with an unstable remission rates ranging from 8% to 100%. Varied characteristics and compliance of enrolled patients might explain this wide range. Considering this, idetification of factors favoring the use of enteral nutrition would be helpful to select preferred patients suitable for enteral nutrition.

In this study, we will observe the role of enteral nutrition in active adult CD. The age, gender, serum CRP, albumin, fecal calprotectin, nutritional risk screening 2002 (NRS2002), involved intestinal segments and other items will be correlated with the changes of Crohn's disease activity index (Best CDAI) and CRP in order to idetify the factors favoring the use of enteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as active CD based on clinical presentation, endoscopic and pathology results
* Has the willing to receive enteral nutrition

Exclusion Criteria:

* No exposure to Glucosteroids or immunosuppressions
* Complete intestinal obstruction

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Active crohn's disease patients from the clinics and wards in the Second Affiliated Hospital, Zhejiang University
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Changes of Best CDAI | 2 months

SECONDARY OUTCOMES:
Changes of serum CRP | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China